CLINICAL TRIAL: NCT06421857
Title: Bipolar Coagulation Versus Suturing During Laparoscopic Endometriotic Cystectomy
Brief Title: Hemostatic Measures During Laparoscopic Cystectomy for Endometrioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Nagat Hesham Abdelhai Mohammed, postgraduate student, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ASU Hemostasis
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Endometrioma
MeSH Terms: conditions — Endometriosis | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suturing (Active Comparator): after ovarian cystectomy for endometrioma, separate sutures were applied if there was significant bleeding
  Interventions: Procedure: suturing
- bipolar electrocoagulation (Active Comparator): after ovarian cystectomy for endometrioma, the inner wall was coagulated using bipolar electrocoagulation if there was significant bleeding
  Interventions: Procedure: bipolar electrocoagulation

INTERVENTIONS:
Procedure: suturing — laparoscopic cystectomy for endometrioma and hemostasis was done using suturing
  Arms: suturing
Procedure: bipolar electrocoagulation — laparoscopic cystectomy for endometrioma and hemostasis was done bipolar electrocoagulation
  Arms: bipolar electrocoagulation

SUMMARY:
laparoscopic excision of ovarian endometriotic cysts is generally recommended because it has been associated with a higher spontaneous conception rate, residual ovarian function after the procedure may be affected

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years
* unilateral endometriotic cyst

Exclusion Criteria:

anovulatory women women with decreased ovarian reserve women receiving hormonal treatment three months prior to surgery women with any contraindication to laparoscopy women with previous ovarian surgery possible ovarian malignancy.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
ovarian reserve | 6 weeks after procedure
  measuring AMH level

CONTACTS AND LOCATIONS:
Overall Officials: Osama Kamel, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No